CLINICAL TRIAL: NCT00081471
Title: A Randomized, Open-label Study of the Effect of Subcutaneous Mircera on Hemoglobin Level/Correction in Non-dialysis Patients With Chronic Kidney Disease
Brief Title: A Study of Mircera in the Treatment of Anemia in Patients With Chronic Kidney Disease Not on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA16738
Record Dates: First submitted 2004-04-13; First posted 2004-04-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa; continuous erythropoietin receptor activator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- 2 (Active Comparator)
  Interventions: Drug: darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa — 0.45 micrograms/kg sc (starting dose) weekly
  Arms: 2
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 0.6 micrograms/kg sc (starting dose) once every 2 weeks
  Arms: 1

SUMMARY:
This study will assess the efficacy and safety of subcutaneous Mircera in the treatment of renal anemia in patients with chronic kidney disease who are not on dialysis and not receiving epoetin or any other erythropoietic substance. The anticipated time on study treatment is 1-2 years and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* chronic kidney disease;
* anemia;
* not on dialysis therapy;
* not receiving epoetin.

Exclusion Criteria:

* women who are pregnant, breastfeeding or using unreliable birth control methods;
* administration of another investigational drug within 4 weeks before screening, or during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2004-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Hemoglobin response rate | Weeks 1-28

SECONDARY OUTCOMES:
Hb concentration over time, time to target Hb response, incidence of RBC transfusions. Vital signs, ECG, adverse events, laboratory values\n\n | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (90):
- United States (21):
  - Los Angeles, California
  - Mather, California
  - Stanford, California
  - Stamford, Connecticut
  - Bay Pines, Florida
  - Ocala, Florida
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - Flushing, New York
  - Cincinnati, Ohio
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Columbia, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Burlington, Vermont
  - Salem, Virginia
  - Morgantown, West Virginia
- Australia (4):
  - Clayton
  - Liverpool
  - Parkville
  - Perth
- Belgium (2):
  - Antwerp
  - Leuven
- Canada (13):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Kamloops, British Columbia
  - New Westminster, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Kitchener, Ontario
  - London, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Saskatoon, Saskatchewan
- France (12):
  - Angers
  - Besançon
  - Chartres
  - Colmar
  - Lille
  - Lyon
  - Nantes
  - Paris
  - Perpignan
  - Salouël
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (6):
  - Aschaffenburg
  - Berlin
  - Bonn
  - Dortmund
  - Düsseldorf
  - Tübingen
- Greece (5):
  - Alexandroupoli
  - Athens
  - Ioannina
  - Piraeus
  - Thessaloniki
- Italy (12):
  - Cagliari
  - Cuneo
  - Genova
  - Lecco
  - Lodi
  - Modena
  - Napoli
  - Padua
  - Pavia
  - Prato
  - Reggio Calabria
  - Roma
- Netherlands (2):
  - Amersfoort
  - Heerlen
- San Juan, Puerto Rico
- Spain (6):
  - Almería
  - Barcelona
  - Lleida
  - Madrid
  - Palma de Mallorca
  - Valencia
- Sweden (2):
  - Borås
  - Umeå
- United Kingdom (4):
  - Birmingham
  - Carshalton
  - Leicester
  - London

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280